CLINICAL TRIAL: NCT00971230
Title: A Pilot Study of Pre-Exposure Prophylaxis (PrEP) to Evaluate Safety, Acceptability, and Adherence in At-risk Populations in Kenya, Africa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Responsible Party: Patricia Fast MD PhD, Chief Medical Officer, International AIDS Vaccine Initiative
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI E001
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
Keywords: HIV; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- FTC/TDF- Daily (Experimental): FTC/TDF dosed daily
  Interventions: Drug: FTC/TDF
- FTC/TDF-Intermittent (Experimental): FTC/TDF dosed intermittently
  Interventions: Drug: FTC/TDF
- Placebo-Daily (Placebo Comparator): Placebo dosed daily
  Interventions: Drug: Placebo
- Placebo-Intermittent (Placebo Comparator): Placebo dosed intermittently
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FTC/TDF — emtricitabine/tenofovir disoproxil fumarate
  Arms: FTC/TDF- Daily; FTC/TDF-Intermittent
Drug: Placebo — Placebo
  Arms: Placebo-Daily; Placebo-Intermittent

SUMMARY:
This study will evaluate the safety and acceptability of an intermittent and daily PrEP regimen using Tenofovir Disoproxil Fumarate plus Emtricitabine (FTC/TDF) in men and women at risk for HIV, and it will directly compare adherence and intracellular drug levels in daily and intermittent PrEP recipients. It will also evaluate the relationship between drug adherence, sexual behavior and intracellular drug levels with an intermittent PrEP regimen. In addition it will evaluate the relationship between adherence to an intermittent PrEP regimen and timing of sexual activity in relation to PrEP dosing. The study will use objective medication event monitoring medication event monitors (MEMS) adherence measurement and evaluate the feasibility of newer adherence measurements such as hair sampling and plasma drug levels. The study will also evaluate the feasibility of using SMS (text messages) to collect sexual activity data in an African setting. It will allow study teams and communities to prepare for potential subsequent larger trials of intermittent PrEP. This study is not sized to evaluate efficacy. If the intermittent PrEP regimen is shown to be safe, feasible in terms of adherence, and achieves intracellular drug levels similar to daily PrEP, these data could be used to design a larger phase 2 study with one or more intermittent PrEP regimens. The goal of such a trial would be to provide bridging data if daily PrEP regimens are found to be effective or to prepare for efficacy or non-inferiority trials of intermittent versus daily PrEP.

Investigation of immune responses associated with FTC/TDF will also be evaluated in the pilot study. The proportion of volunteers on FTC/TDF with HIV-specific immune responses, due to exposures that did not lead to established HIV infection, will be assessed at 2-3 time points and compared to responses in volunteers assigned to placebo. Immune responses may be correlated with risk behavior and host factors, such as human leukocyte antigen (HLA) type. As noted above, very few HIV infections are expected to occur during the study, so correlation of HIV-specific immune responses and protection from infection or attenuation of disease progression will not be possible until a larger study is conducted.

ELIGIBILITY:
Inclusion Criteria

* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study
* Has understood the information provided and has provided written informed consent before any study-related procedures are performed
* Willing to undergo HIV testing, STI screening, HIV counselling and receive HIV and STI test results
* At risk for HIV infection as defined by at least one of the following:

  * Current sexually-transmitted infection (STI) or STI in the previous 3 months
  * In the past 3 months had multiple episodes of unprotected vaginal sex
  * In the past 3 months had multiple episodes of unprotected anal sex
  * In the past 3 months engaged in sex work for money or drugs
* If a female of childbearing potential (i.e., not post-menopausal or surgically sterile), using an effective method of non-barrier contraception (hormonal contraceptive; intrauterine device (IUD); surgical sterility) from 7 days prior to randomization until the end of the study. All female volunteers must be willing to undergo urine pregnancy tests

Exclusion Criteria

* Confirmed HIV-1 or HIV-2 infection
* Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator would make the volunteer unsuitable for the study, including severe infections requiring treatment such as tuberculosis, and alcohol or drug abuse
* Any of the following abnormal laboratory parameters:

  * Haemoglobin <9.0 g/dL
  * Creatinine clearance <80mL/min, as calculated by Cockcroft-Gault equation
  * AST: >2.5 x ULN
  * ALT: >2.5 x ULN
  * Total bilirubin >1.5 x ULN
  * Serum amylase >1.5 x ULN
  * Serum phosphorus <2.4 mg/dL
  * Urinalysis: Two abnormal dipsticks showing any of the following:

    * blood = 2+ or more (not due to menses)
    * protein = 1+ or more
    * leucocytes = 2+ or more
    * glucose= 1+ or more
* Confirmed diagnosis of chronic hepatitis B infection (HBsAg positive)
* If female, pregnant or planning a pregnancy within 4 months after enrolment or lactating
* Participation in another clinical study of an investigational product currently, within the 3 months prior to enrolment or expected participation during this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: The proportion of volunteers with moderate and greater severity clinical adverse events; mild, moderate and greater severity of renal toxicities, and other moderate and severe laboratory abnormalities. | 6 months
Acceptability: The proportion of volunteers who report willingness to use the study regimen | 6 months
Intracellular drug concentrations: The mean intracellular drug concentration for each group assigned to FTC/TDF | 6 months
Adherence: Proportion of volunteers who took, by MEMS data, at least 80% of expected doses of the IP; Proportion of volunteers assigned to FTC/TDF who have detectable drug plasma levels within 48 hrs of use. | 6 months
Behavioral: Reported number of steady and casual sex partners; Frequency of unprotected vaginal and/or anal intercourse; Substance use prior to or during sex | 6 months

SECONDARY OUTCOMES:
Proportion of volunteers who report somewhat high or high levels of burden in using electronic medication monitoring to measure adherence, and using cell phone communication to measure sexual activity | 6 months
The proportion of study days with missing SMS sexual activity data | 6 months
The proportion of volunteers who report sharing medications | 6 months
The proportion of volunteers assigned to placebo who have detectable intracellular drug levels | 6 months
The proportion of volunteers with HIV-specific immune responses as measured by analysis of cellular or humoral immune response, or changes in gene regulation as measured by microarray or proteomic techniques | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaudensia Mutua, MB.ChB, MPH, Principal Investigator — Kenya AIDS Vaccine Initiative, University of Nairobi; E.J. Sanders, MD, MPH, PhD, Principal Investigator — Kenya Medical Research Institute, Center for Geographic Medicine Research - Coast; Omu Anzala, MB.ChB, Phd, Study Chair — Kenya AIDS Vaccine Initiative, University of Nairobi
Locations (2):
- Kenya (2):
  - Kenya Medical Research Institute, Center for Geographic Medicine Research - Coast, Kilifi, Kilifi County
  - Kenya AIDS Vaccine Initiative, University of Nairobi, Nairobi, Nairobi County

REFERENCES:
- [Derived] Baxi SM, Liu A, Bacchetti P, Mutua G, Sanders EJ, Kibengo FM, Haberer JE, Rooney J, Hendrix CW, Anderson PL, Huang Y, Priddy F, Gandhi M. Comparing the novel method of assessing PrEP adherence/exposure using hair samples to other pharmacologic and traditional measures. J Acquir Immune Defic Syndr. 2015 Jan 1;68(1):13-20. doi: 10.1097/QAI.0000000000000386. PMID 25296098
- [Derived] Mutua G, Sanders E, Mugo P, Anzala O, Haberer JE, Bangsberg D, Barin B, Rooney JF, Mark D, Chetty P, Fast P, Priddy FH. Safety and adherence to intermittent pre-exposure prophylaxis (PrEP) for HIV-1 in African men who have sex with men and female sex workers. PLoS One. 2012;7(4):e33103. doi: 10.1371/journal.pone.0033103. Epub 2012 Apr 12. PMID 22511916
- See also: International AIDS Vaccine Initiative — http://www.iavi.org